CLINICAL TRIAL: NCT06439199
Title: Single-center, Biological, Uncontrolled, Prospective Study Evaluating the Dosage of Plasma Cytokines Including the FLT3 (FMS-like Tyrosine Kinase 3) Ligand and IL6 With a View to Making a First Estimate of Their Prognostic Value on the Outcome of Patients Treated With Non-intensive Chemotherapy Such as Azacytidine for Acute Myelogenous Leukemia (AML), High Risk Myelodysplastic Syndrome (HR-MDS) or Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Biological, Prospective Study Evaluating the Dosage of Plasma Cytokines Including the FLT3 Ligand and IL6 of Patients Treated With Non-intensive Chemotherapy
Acronym: CYTOK-AZA
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC23_0332
Record Dates: First submitted 2024-02-09; First posted 2024-06-03 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: Cytokine; IL 6; FLT3 Ligand; AML; CMML; HR MDS; Azacytidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the weekly blood samples taken in the day hospital as part of the treatment, an additional 9 ml EDTA tube will be taken, during the first 2 cycles for group 1 and during the first 3 cycles for group 2.This additional tube will be used to supply this biocollection and to promote the development of knowledge in the field of acute myeloidblastic leukemia, myelodysplasia and chronic myelomonocytic leukemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Azacytidine and Venetoclax: 40 patients treated with Azacytidine and Venetoclax +/- another molecule according to the following schedule:
  * Azacytidine 75 mg/m² D1 to D7 SC
  * Venetoclax: 400 mg/day orally in 1 dose between 14 and 28 days per cycle. The cycles will be 28 days long and will be carried out until relapse or death. Cytokine assays will be carried out on D1, D8, D15 and D22 of each cycle for 2 cycles.
- Azacytidine: 20 patients treated with Azacytidine +/- another molecule according to the following schedule:
  • Azacytidine 75 mg/m² D1 to D7 SC The cycles will be 28 days long and will be carried out until relapse or death. The cytokine assays will be carried out on D1, D8, D15 and D22 of each cycle for 3 cycles.
  The duration of follow-up for a patient is 12 months from day 1 of the first cycle.

SUMMARY:
There are 2 possible treatments for the treatment of Acute Myelogenous Leukemia (AML), high-risk myelodysplastic syndromes (HR-MDS) or chronic myelomonocytic leukemia (CMML): intensive curative chemotherapy , and for over-aged or co-morbid patients , non-intensive palliative chemotherapy with a hypomethylating agent (Azacytidine) associated or not with venetoclax.

Pro-inflammatory cytokines and in particular IL-6 (Interleukin 6) seem to play a key role in the chemoresistance of solid cancers and AML : it would be associated with a poor prognosis of AML , would promote the proliferation of leukemic blasts , and would promote the progression of MDS to AML .

In AML treated with intensive chemotherapy, researchers demonstrated that a particular kinetic profile of the FLT3 ligand and IL6 at day 22 could very significantly predict the survival of patients with AML .

It therefore seems interesting to study the plasma cytokine profiles in patients with AML, HR-MDS or CMML treated non-intensively, and to see if researchers observe the same prognostic correlation as during intensive chemotherapy.

DETAILED DESCRIPTION:
Patients will be divided into 2 groups treated according to a non-intensive chemotherapy :

Group 1 : 40 patients treated with Azacytidine and Venetoclax +/- another molecule according to the following schedule:

* Azacytidine 75 mg/m² D1 to D7 SC
* Venetoclax: 400 mg/day orally in 1 dose between 14 and 28 days per cycle. The cycles will be 28 days long and will be carried out until relapse or death. Cytokine assays will be carried out on D1, D8, D15 and D22 of each cycle for 2 cycles.

Group 2 : 20 patients treated with Azacytidine +/- another molecule according to the following schedule:

• Azacytidine 75 mg/m² D1 to D7 SC The cycles will be 28 days long and will be carried out until relapse or death. The cytokine assays will be carried out on D1, D8, D15 and D22 of each cycle for 3 cycles.

The duration of follow-up for a patient is 12 months from day 1 of the first cycle.

ELIGIBILITY:
Inclusion Criteria :

* Age >=18 years
* AML or SMD-HR or CMML in first line or in relapse receiving a hypomethylating agent +/- another molecule or a hypomethylating agent in combination with venetoclax +/- another molecule.
* Patient having agreed to participate in the study (information note signature) and having signed the biocollection consent

Exclusion Criteria :

* No social security or any other regime
* Pregnant women or patient unable to take contraception in case of fertility
* Breastfeeding women
* Minors
* Adults under guardianship, curators or safeguard of justice

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 patients treated with Azacytidine and Venetoclax +/- another molecule and 20 patients treated with Azacytidine +/- another molecule.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of cytokine profiles (Flt3-L, IL (Interleukin) 1beta, IL6, IL8/CXCL8, IL10, IL15, IL17A, IL17E, IL17-F, IL18, GM-CSF, TNFalpha) in patients treated non-intensively for AML, SMD-HR or an LMMC. | 2 years
  Determination of plasma cytokines (Flt3-L, IL1beta, IL6, IL8/CXCL8, IL10, IL15, IL17A, IL17E, IL17-F, IL18, GM-CSF (granulocyte-monocyte colony-stimulating factor, TNFalpha) by Luminex at diagnosis and during treatment of adult patients with of AML, SMD-HR (High risk myelodysplastic syndrome) or CMML(Chronic myelomonocytic leukemia) treated non-intensively

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No